CLINICAL TRIAL: NCT01778608
Title: Feasibility Test of a Handset Device to Detect Sedation Levels and Loss of Consciousness During Propofol Administration
Brief Title: Feasability Test of a Handset Device to Detect Levels of Sedation and Loss of Consciousness
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: PCS-001
Record Dates: First submitted 2012-05-31; First posted 2013-01-29 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Conscious Sedation
Keywords: Sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sedation is often administered to relieve anxiety and discomfort during uncomfortable procedures in elderly patients. Patient control of sedation offers many potential benefits for patients and healthcare professionals, including improved safety and patient satisfaction. The investigators overall goal is to develop a patient controlled intravenous sedation system that is effective but very safe for the patient, and requires minimal supervision by a doctor or nurse. To fulfill these criteria, a sedation system should incorporate fail-safe safety mechanisms. A key safety-critical component is a method of objectively assessing the degree of sedation of the patient, and of preventing him from self-administering unsafe doses of the sedative drug. The investigators have designed a new sedation system that uses a measure of the speed of response of the patient to a defined non-noxious stimulus to determine whether or not it is safe to allow him to self-administer further levels of sedation. Before being able to execute a volunteer study in order to determine a rational selection of optimal threshold response time, a feasibility test on the handset device is required.

ELIGIBILITY:
Inclusion Criteria:

* age 50-72 years

Exclusion Criteria:

* volunteer refusal
* patient age >72 years
* significant cardiovascular or respiratory disease
* latex allergy

Ages: 50 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients requiring anaesthesia for clinical surgical care. ASA physical status I, II or III
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Response times | Continuously shortly before (baseline)
  Response time between non-noxious stimulus and activation of handset device
response time | during induction of anesthesia
  Response time between non-noxious stimulus and activation of handset device

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands